CLINICAL TRIAL: NCT00770146
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of ISIS 301012 (Mipomersen) as Add-on Therapy in High Risk Hypercholesterolemic Patients
Brief Title: Safety and Efficacy of Mipomersen (ISIS 301012) As Add-on Therapy in High Risk Hypercholesterolemic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 301012-CS12
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2013-03-20 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection once a week for 26 weeks.
  Interventions: Drug: Placebo
- Mipomersen (Experimental): Participants received mipomersen 200 mg as a subcutaneous injection once a week for 26 weeks.
  Interventions: Drug: Mipomersen sodium

INTERVENTIONS:
Drug: Mipomersen sodium — 200 mg/mL
  Other Names: ISIS 301012; Kynamro™
  Arms: Mipomersen
Drug: Placebo — 1 mL matching placebo (i.e., vehicle consisting of 9 mg of sodium chloride, 0.004 mg of riboflavin, filled to 1 mL with water).
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of dosing with mipomersen for 26 weeks in patients with high cholesterol who are on a maximally tolerated dose of statin and who have a diagnosis that puts them at least at high risk of coronary heart disease (CHD).

DETAILED DESCRIPTION:
Hypercholesterolemia is characterized by markedly elevated low density lipoproteins (LDL). Elevated LDL is a major risk factor for CHD.

Mipomersen is an antisense drug that reduces a protein in the liver cells called apolipoprotein B (apo-B). Apo-B plays a role in producing low density lipoprotein cholesterol (LDL-C) (the "bad" cholesterol) and moving it from the liver to one's bloodstream. High LDL-C is an independent risk factor for the development of CHD or other diseases of blood vessels. It has been shown that lowering LDL-C reduces the risk of heart attacks and other major adverse cardiovascular events. The purpose of this study is to determine whether mipomersen safely and effectively lowers LDL-C in patients with high cholesterol who are at high risk for CHD and who are already on the maximally tolerated dose of statin.

This study consisted of a 26-week treatment period and a 24-week post-treatment follow-up period. Participants who finished treatment or who discontinued prematurely from the study for any reason were assessed for safety for 24 weeks after the last study drug dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypercholesterolemia (LDL-C ≥ 100 mg/dL)
* At high risk of CHD
* On stable, maximally tolerated statin therapy for 8 weeks
* On stable, low fat diet for 12 weeks
* Stable weight for 6 weeks

Exclusion Criteria:

* Significant health problems in the recent past including heart attack, stroke, coronary syndrome, unstable angina, heart failure, significant arrhythmia, hypertension, liver disease, cancer, type I diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (54):
- United States (54):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Muscle Shoals, Alabama
  - Litchfield Park, Arizona
  - Beverly Hills, California
  - Escondido, California
  - Los Angeles, California
  - Mission Viejo, California
  - Newport Beach, California
  - San Diego, California
  - Santa Rosa, California
  - Thousand Oaks, California
  - Westlake Village, California
  - Aventura, Florida
  - Inverness, Florida
  - Jacksonville, Florida
  - Longwood, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Pembroke Pines, Florida
  - Pensacola, Florida
  - Ponte Verda, Florida
  - Port Orange, Florida
  - Sandy Springs, Georgia
  - Chicago, Illinois
  - Bloomingtom, Indiana
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Brockton, Massachusetts
  - New Bedford, Massachusetts
  - Edina, Minnesota
  - Kansas City, Missouri
  - Berlin, New Jersey
  - Johnson City, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Wilson, North Carolina
  - Cincinnati, Ohio
  - Mentor, Ohio
  - Norman, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Lansdale, Pennsylvania
  - Murrells Inlet, South Carolina
  - Simpsonville, South Carolina
  - Spartanburg, South Carolina
  - Rapid City, South Dakota
  - Dallas, Texas
  - Grapevine, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Olympia, Washington

REFERENCES:
- [Derived] Santos RD, Raal FJ, Catapano AL, Witztum JL, Steinhagen-Thiessen E, Tsimikas S. Mipomersen, an antisense oligonucleotide to apolipoprotein B-100, reduces lipoprotein(a) in various populations with hypercholesterolemia: results of 4 phase III trials. Arterioscler Thromb Vasc Biol. 2015 Mar;35(3):689-99. doi: 10.1161/ATVBAHA.114.304549. Epub 2015 Jan 22. PMID 25614280
- [Derived] Thomas GS, Cromwell WC, Ali S, Chin W, Flaim JD, Davidson M. Mipomersen, an apolipoprotein B synthesis inhibitor, reduces atherogenic lipoproteins in patients with severe hypercholesterolemia at high cardiovascular risk: a randomized, double-blind, placebo-controlled trial. J Am Coll Cardiol. 2013 Dec 10;62(23):2178-84. doi: 10.1016/j.jacc.2013.07.081. Epub 2013 Sep 4. PMID 24013058

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five hundred and seventy-seven patients were screened and 158 patients were randomized at 43 study centers in a 2:1 ratio to receive mipomersen or placebo once a week for 26 weeks. Participants who finished treatment or who discontinued prematurely from the study for any reason were assessed for safety for 24 weeks after the last study drug dose.
Period: Treatment Period
Arm/Group | Placebo | Mipomersen
Started | 53 | 105
Treated | 52 | 105
Full Analysis Set | 50 (Treated patients with a valid baseline & post-baseline LDL-C measurement) | 101 (Treated patients with a valid baseline & post-baseline LDL-C measurement)
Completed | 44 | 60
Not Completed | 9 | 45
Not completed — Withdrawal by Subject | 6 | 13
Not completed — Adverse Event | 2 | 26
Not completed — Other | 1 | 5
Not completed — Protocol non-compliance | 0 | 1
Period: Follow-up Period
Arm/Group | Placebo | Mipomersen
Started | 53 | 105
Completed | 42 | 85
Not Completed | 11 | 20
Not completed — Withdrawal by Subject | 7 | 13
Not completed — Adverse Event | 0 | 2
Not completed — Other | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mipomersen | Total
Number analyzed (Participants) | 52 | 105 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline data are provided for the Safety Set.
  years | 59.3 (9.5) | 59.3 (10.0) | 59.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 53 | 76
  Male | 29 | 52 | 81
Race/Ethnicity, Customized [Number; unit: participants]
  White | 40 | 83 | 123
  Black | 11 | 20 | 31
  American Indian or Alaskan Native | 1 | 1 | 2
  Other race | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 9 | 16 | 25
  Not Hispanic or Latino | 43 | 89 | 132
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (4.42) | 30.7 (4.61) | 30.4 (4.55)
Waist/hip ratio [Mean (Standard Deviation); unit: ratio] | 0.94 (0.07) | 0.94 (0.06) | 0.94 (0.06)
Metabolic syndrome [Number; unit: participants] — A patient was classified as having metabolic syndrome if any 3 of the following risk factors existed: 1) Waist circumference ≥102 cm (men) or ≥88 cm (women); 2) Triglycerides ≥150 mg/dL*; 3) High density lipoprotein cholesterol <40 mg/dL (men) or <50 mg/dL (women)*; 4) Systolic blood pressure ≥130 or diastolic ≥85 mmHg *; 5) Fasting glucose ≥100 mg/dL *.
  * = or on medication for the specified risk factor.
  participants
    No | 12 | 32 | 44
    Yes | 40 | 73 | 113
Tobacco use [Number; unit: participants]
  Current | 11 | 18 | 29
  Non-current | 19 | 31 | 50
  Never | 22 | 56 | 78
Alcohol use [Number; unit: participants]
  Current | 20 | 50 | 70
  Non-current | 12 | 24 | 36
  Never | 20 | 31 | 51
Diabetic status at screening [Number; unit: participants]
  Yes | 30 | 58 | 88
  No | 22 | 47 | 69
Cardiovascular history [Number; unit: participants] — Participants may be counted in more than one category.
  participants
    Angina | 5 | 9 | 14
    Coronary heart disease (CHD) | 21 | 52 | 73
    Myocardial infarction | 11 | 17 | 28
    Coronary artery bypass graft surgery | 4 | 14 | 18
    Percutaneous coronary intervention | 4 | 18 | 22
    Coronary artery disease without event | 6 | 14 | 20
    Other clinical atherosclerotic disease | 3 | 11 | 14
    Peripheral artery disease | 1 | 5 | 6
    Abdominal aortic aneurysm | 1 | 0 | 1
    Carotid | 1 | 8 | 9
    CHD or other atherosclerotic disease | 24 | 58 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at the Primary Efficacy Time Point
Description: LDL cholesterol was measured in mg/dL. Samples were taken following an overnight fast. LDL-C was obtained using Friedewald's calculation for patients with triglycerides ≤400 mg/dL and was directly measured by the central laboratory using ultracentrifugation for patients with triglycerides >400 mg/dL. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: Baseline (the average of the screening and Day 1 pre-treatment assessments) and the Primary Efficacy Time point (PET; Week 28 or the post-baseline visit closest to 14 days after the last dose).
Population: The Full Analysis Set, which consisted of all randomized patients who received at least 1 injection of study drug (mipomersen or placebo) and with a valid baseline and at least 1 post-baseline LDL-C measurement.
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
percentage of baseline | -3.4 (24.22) [-14.8 to 11.8] | -40.2 (26.85) [-56.4 to -19.1]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Based upon prior clinical study experience with mipomersen, it was estimated that the standard deviation of the percent change in LDL-C is approximately 22%. With at least 20 patients in the control group and 40 patients in the mipomersen-treated group, this study would have at least 90% power to detect a 20% difference between the 2 groups; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Statistical significance was concluded if p ≤ 0.05

2. Primary Outcome: Low-density Lipoprotein Cholesterol (LDL-C) at Baseline and at the Primary Efficacy Time Point
Description: The primary efficacy time point (PET) was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
mg/dL
  Baseline | 112 (38.6) [101 to 134] | 116 (31.7) [106 to 137]
  Primary efficacy time point | 109 (35.1) [90 to 128] | 69 (32.4) [51 to 98]

3. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Primary Efficacy Time Point
Description: Apolipoprotein B was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
percentage of baseline | -1.7 (18.09) [-12.6 to 7.5] | -40.6 (23.59) [-53.9 to -22.6]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Inflation of type 1 error was controlled by specifying a small number of secondary parameters and a sequential inferential approach in which inferential conclusions about each successive parameter required statistical significance of the prior one

4. Secondary Outcome: Apolipoprotein B at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
mg/dL
  Baseline | 106 (30.1) [98 to 132] | 114 (25.2) [102 to 129]
  Primary efficacy time point | 108 (27.2) [91 to 122] | 64 (30.7) [52 to 95]

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at the Primary Efficacy Time Point
Description: Total cholesterol was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
percentage of baseline | -2.7 (14.58) | -26.4 (18.65)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Total Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
mg/dL
  Baseline | 200.0 (42.1) | 202.6 (36.8)
  Primary efficacy time point | 192.2 (38.3) | 147.4 (39.9)

7. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol at the Primary Efficacy Time Point
Description: Non-high-density lipoprotein cholesterol was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
percentage of baseline | -1.2 (20.43) [-13.6 to 11.5] | -38.7 (23.75) [-54.0 to -24.2]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]

8. Secondary Outcome: Non-High-Density Lipoprotein Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
mg/dL
  Baseline | 144 (44.4) [125 to 175] | 144 (35.1) [132 to 171]
  Primary efficacy time point | 140 (38.7) [115 to 165] | 90 (38.3) [67 to 116]

9. Other Pre Specified Outcome: Percent Change From Baseline in Triglycerides at the Primary Efficacy Time Point
Description: Triglycerides were measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
percentage of baseline | 2.7 (53.26) [-24.0 to 24.2] | -26.2 (29.21) [-48.1 to -8.8]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustments were made for tertiary parameters

10. Other Pre Specified Outcome: Triglycerides at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
mg/dL
  Baseline | 139 (66.1) [98 to 176] | 143 (65.3) [105 to 175]
  Primary efficacy time point | 135 (97.5) [96 to 177] | 88 (55.7) [67 to 128]

11. Other Pre Specified Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at the Primary Efficacy Time Point
Description: High-density lipoprotein cholesterol (HDL-C) was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
percentage of baseline | 2.2 (16.44) | 2.2 (17.99)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.977, t-test, 2 sided — No adjustments were made for tertiary parameters

12. Other Pre Specified Outcome: High-Density Lipoprotein Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
mg/dL
  Baseline | 48.4 (15.9) | 50.8 (12.0)
  Primary efficacy time point | 48.9 (16.1) | 51.1 (12.3)

13. Other Pre Specified Outcome: Percent Change From Baseline in Lipoprotein (a) at the Primary Efficacy Time Point
Description: Lipoprotein (a) was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
percentage of baseline | 2.3 (28.09) | -24.0 (24.47)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — No adjustments were made for tertiary parameters

14. Other Pre Specified Outcome: Lipoprotein (a) at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
mg/dL
  Baseline | 51.1 (48.6) | 54.3 (57.0)
  Primary efficacy time point | 49.5 (47.3) | 39.6 (47.0)

15. Other Pre Specified Outcome: Percent Change From Baseline in Very Low Density Lipoprotein Cholesterol at the Primary Efficacy Time Point
Description: Very low density lipoprotein (VLDL) cholesterol was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
percentage of baseline | 1.9 (53.83) [-23.1 to 26.3] | -26.7 (28.75) [-46.8 to -9.1]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustments were made for tertiary parameters

16. Other Pre Specified Outcome: Very Low Density Lipoprotein Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
mg/dL
  Baseline | 28 (13.2) [20 to 35] | 29 (12.1) [21 to 35]
  Primary efficacy time point | 27 (16.3) [19 to 35] | 18 (11.1) [13 to 26]

17. Other Pre Specified Outcome: Percent Change From Baseline in the Ratio of LDL Cholesterol to HDL Cholesterol at the Primary Efficacy Time Point
Description: The ratio of low-density lipoprotein (LDL) cholesterol to high-density lipoprotein (HDL) cholesterol was measured at Baseline and the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
percentage of baseline | -5.3 (25.31) | -37.4 (27.24)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — No adjustments were made for tertiary parameters

18. Other Pre Specified Outcome: Ratio of LDL Cholesterol to HDL Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
ratio
  Baseline | 2.82 (1.383) | 2.54 (0.854)
  Primary efficacy time point | 2.54 (1.147) | 1.54 (0.761)

19. Other Pre Specified Outcome: Percent Change From Baseline in Apolipoprotein A1 at the Primary Efficacy Time Point
Description: Apolipoprotein A1 was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
percentage of baseline | -1.0 (11.16) | -5.6 (12.56)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.032, t-test, 2 sided — No adjustments were made for tertiary parameters

20. Other Pre Specified Outcome: Apolipoprotein A1 at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 50 | 101
mg/dL
  Baseline | 150.8 (30.5) | 156.8 (25.4)
  Primary efficacy time point | 147.8 (27.3) | 146.8 (24.5)

ADVERSE EVENTS:
Time Frame: Up to Week 28 (2 weeks after last dose)
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Placebo | Mipomersen
Serious Adverse Events (participants affected / at risk) | 4/52 | 7/105
Other Adverse Events (participants affected / at risk) | 42/52 | 97/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | Mipomersen (N=105)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Electrocardiogram abnormal (Investigations) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | Mipomersen (N=105)
Anaemia (Blood and lymphatic system disorders) | 1 | 5
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac discomfort (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 4
Tachycardia (Cardiac disorders) | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Adrenal mass (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Blepharitis (Eye disorders) | 0 | 1
Cataract nuclear (Eye disorders) | 0 | 1
Ectropion (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Keratopathy (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Diverticulum (Gastrointestinal disorders) | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 11
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 2
Pancreatic atrophy (Gastrointestinal disorders) | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 1
Pancreatic duct dilatation (Gastrointestinal disorders) | 2 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4
Asthenia (General disorders) | 0 | 2
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 0 | 8
Fatigue (General disorders) | 4 | 13
Feeling jittery (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 7
Injection site discolouration (General disorders) | 2 | 19
Injection site discomfort (General disorders) | 1 | 2
Injection site dryness (General disorders) | 0 | 1
Injection site erythema (General disorders) | 2 | 56
Injection site exfoliation (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 3 | 17
Injection site haemorrhage (General disorders) | 1 | 6
Injection site induration (General disorders) | 0 | 5
Injection site inflammation (General disorders) | 0 | 2
Injection site nodule (General disorders) | 4 | 13
Injection site oedema (General disorders) | 0 | 6
Injection site pain (General disorders) | 11 | 57
Injection site pallor (General disorders) | 0 | 1
Injection site papule (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 0 | 31
Injection site rash (General disorders) | 0 | 6
Injection site reaction (General disorders) | 0 | 5
Injection site recall reaction (General disorders) | 0 | 2
Injection site swelling (General disorders) | 0 | 17
Injection site urticaria (General disorders) | 0 | 3
Injection site vesicles (General disorders) | 0 | 5
Injection site warmth (General disorders) | 0 | 9
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 3
Pain (General disorders) | 1 | 6
Pyrexia (General disorders) | 3 | 5
Vessel puncture site haemorrhage (General disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 3 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 11
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 4
Acarodermatitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 2
Cellulitis (Infections and infestations) | 0 | 1
Conjunctivitis viral (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 6
Labyrinthitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 6
Oral herpes (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 4
Tinea pedis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 10
Urinary tract infection (Infections and infestations) | 5 | 12
Viral infection (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 9
Aspartate aminotransferase increased (Investigations) | 1 | 5
Beta 2 microglobulin urine increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 2 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood testosterone decreased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 2 | 0
Body temperature increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Eosinophil percentage increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 0 | 1
Helicobacter test positive (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 4
International normalised ratio increased (Investigations) | 1 | 2
Liver function test abnormal (Investigations) | 0 | 8
Platelet count decreased (Investigations) | 0 | 1
Protein urine present (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 1
QRS axis abnormal (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 9
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 5
Headache (Nervous system disorders) | 3 | 10
Hyporeflexia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 2
Mental impairment (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 3
Claustrophobia (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 3
Disorientation (Psychiatric disorders) | 0 | 1
Dysphoria (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 5
Libido decreased (Psychiatric disorders) | 1 | 0
Listless (Psychiatric disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 3
Endometrial atrophy (Reproductive system and breast disorders) | 0 | 1
Genital lesion (Reproductive system and breast disorders) | 0 | 1
Premenstrual syndrome (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal turbinate abnormality (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 3 | 11
Hypotension (Vascular disorders) | 0 | 2
Intermittent claudication (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study the PI may publish the results of his/her data from the study. The PI shall provide the sponsor with an advance copy at least 60 days prior to planned submission and the Sponsor shall have 60 days to review (contracts have variable timeframes; maximum times are stated here). The sponsor may request the deletion of any confidential information, or a delay in submission for an additional period not to exceed 90 days.